CLINICAL TRIAL: NCT04245241
Title: Effects of High-Flow Nasal Cannula Therapy on Lung Recruitment and Lung Strain Change Assessed by Electrical Impedance Tomography
Brief Title: Effects of High-Flow Nasal Cannula Therapy Assessed by Electrical Impedance Tomography
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EIT-HFNC
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: High-flow Nasal Cannula; Electrical Impedance Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: High-flow nasal cannula (HFNC) — 24 patients who receiving HFNC within 24 hours after extubation were prospectively enrolled in this study. EIT was used to monitor regional lung ventilation distributions at baseline (conventional oxygen therapy) and three flow rate levels of HFNC therapy (20, 40 and 60 L/min).

SUMMARY:
This study aimed to determine the effects of HFNC therapy on lung recruitment and lung strain change assessed by electrical impedance tomography (EIT)

ELIGIBILITY:
* Inclusion Criteria:
* Patient who received a HENC therapy within 24 h after the extubation

Exclusion Criteria:

* Aged <18 years
* Pregnancy
* Body mass index (BMI) over 50 kg/m2
* ribcage malformation .any contraindication of using EIT monitoring (automatic implantable cardioverter defibrillator, chest skin injury, etc.).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult critically ill patients, who received a HENC therapy within 24 h after the extubation, were enrolled.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
lung regional ventilation distribution | minute 80
  lung regional ventilation distribution measured by EIT

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Peking Union Medical College Hospital, Peking Union Medical College, Chinese Academy of Medical Sciences,, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang R, He H, Yun L, Zhou X, Wang X, Chi Y, Yuan S, Zhao Z. Effect of postextubation high-flow nasal cannula therapy on lung recruitment and overdistension in high-risk patient. Crit Care. 2020 Mar 6;24(1):82. doi: 10.1186/s13054-020-2809-7. PMID 32143664